CLINICAL TRIAL: NCT02408029
Title: Trauma Equivalency Study of the CORA® and TEG® 5000 Systems
Status: Completed | Type: Observational
Sponsor: Coramed Technologies LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 01-229
Record Dates: First submitted 2015-03-25; First posted 2015-04-03 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Trauma
Keywords: Focus; Testing Performance; CORA Hemostasis System
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trauma Patients Group: Patients undergoing treatment for injuries and trauma.
  Interventions: Other: Observational study - no intervention

INTERVENTIONS:
Other: Observational study - no intervention

SUMMARY:
This study is being performed to obtain data about the CORA System when used in a trauma clinical setting. The CORA analyzer is a new device that is currently being tested in trauma clinical applications and is not yet cleared for this purpose by the Food and Drug Administration (FDA) for sale in the United States.

DETAILED DESCRIPTION:
The purpose of the study is to validate the CORA System by comparing the results of this test to that of the standard of care device called the TEG 5000 system. Both systems evaluate hemostasis, a highly complex and interactive process involving many protein and cellular elements, especially platelets, occurring in a series of interrelated phases, which results in either normal hemostasis or a tendency toward bleeding or clotting complications.

The study protocol specifies testing using multiple reagents which are similar for both the CORA and TG 5000 systems. Tests are run in duplicate on blood samples taken from patients undergoing treatment for injuries and trauma. Following the protocol defined in CLSI Standard EP09-A2, equivalence between the two systems will be demonstrated if the conclusions from the Standard Section 7, Interpreting Results and Comparing to Internal Performance Criteria, are found to be acceptable.

All blood samples drawn for this study will use venous blood. Only citrated or heparinized whole blood samples are used. All samples are tested twice (run in duplicate). Quality Control procedures are run on both instruments at a frequency specified by the manufacturers. Results obtained from this testing are not used to make treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Complete patient history including age, race, gender and type of trauma should be documented

Exclusion Criteria:

* Patients under the age of 18
* Native whole blood will not be used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or over undergoing care for trauma.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Composite measure: Blood coagulation and hemostasis parameters R (min), C-ACT (min), K (min), Angle (degrees), MA (mm) and LY30 (%) parameters for both TEG 5000 and CORA systems | 1 day, measured at time of trauma treatment; no follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Charles E Wade, Ph.D., Principal Investigator — The University of Texas Health Science Center, Houston; Martin A Schreiber, M.D., Principal Investigator — Oregon Health and Science University; Mark Walsh, M.D., Principal Investigator — Indiana School of Medicine, South Bend Notre Dame Campus
Locations (3):
- United States (3):
  - Indiana School of Medicine South Bend Notre Dame Campus, South Bend, Indiana
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas Health Science Center at Houston, Houston, Texas